CLINICAL TRIAL: NCT04203290
Title: Comparison of General Anesthesia and Combined General Thoracic Epidural Anesthesia on End Tidal Volatile Anesthetic Concentration in Cases Which Depth of Anesthesia is Adjusted Using Entropy Monitoring; A Prospective Trial
Brief Title: End Tidal Anesthetic Concentration in Different Anesthesia Techniques Where Depth of Anesthesia Adjusted With Entropy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nuzhet Mert Senturk, MD, Prof, Professor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2018/1377
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: General Anesthesia; Inhalation; Gas
Keywords: Minumum alveoler concentration; Entropy monitorining; General anesthesia; General anesthesia combined with TEA
MeSH Terms: conditions — Respiratory Aspiration; Mucopolysaccharidosis IV | interventions — Bupivacaine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia (Active Comparator): Patients will be applyed 0.03 mg/kg midazolam, 2 mcg/kg fentanyl, propofol until reaching the appropriate anesthetic depth by observing entropy value (40-60) and 0.5 mg/kg rocuronium for anesthesia induction, after intubation sevoflurane will be used for anesthesia maintenance with low flow anesthesia (0.5 l/min).
  Interventions: Drug: Sevoflurane
- General anesthesia combined with thoracic epidural anesthesia (Active Comparator): Before anesthesia induction epidural catheter will be inserted giving 7 ml bupivacaine %0.25 in saline + 50 mcg fentanyl after confirming the location of catheter, following 15 minutes the standard anesthesia induction will be applied ( 0.03 mg/kg midazolam, 2 mcg/kg fentanyl, propofol until reaching the appropriate anesthetic depth by observing entropy value (40-60) and 0.5 mg/kg rocuronium ). For anesthesia maintenance epidural infusion will be applied ( 7ml/h %0.25 bupivacaine solution) together with low flow (0.5 l/min) sevoflurane anesthesia.
  Interventions: Drug: Bupivacaine; Drug: Sevoflurane

INTERVENTIONS:
Drug: Bupivacaine — %0.25 bupivacaine solution
  Other Names: marcaine
  Arms: General anesthesia combined with thoracic epidural anesthesia
Drug: Sevoflurane — End tidal sevoflurane concentration
  Other Names: Sevorane

SUMMARY:
The aim of this study is to adjust the end tidal inhalation anesthetic concentration by observing the entropy value in patients who will be provided anesthesia maintenance with volatile anesthetics after applying the routine epidural anesthesia technique and to observe the end tidal volatile concentration that will provide to remain in the target entropy limits during the operation.

DETAILED DESCRIPTION:
The hypothesis of this study is that in general anesthesia cases which is combined with thoracic epidural anesthesia (TEA), lower alveolar concentration will be required to reach the same anesthesia depth. The main aim of the study is observing and comparing the alveolar concentrations of anesthetic agents with entropy monitoring which is an anesthesia depth monitor in major abdominal surgeries where general anesthesia is combined or not with TEA.

In cases where TEA is combined with general anesthesia or not, anesthesia depth will be effectively monitored by entropy monitoring, in this way the adequate depth of anesthesia will be provided with the use of minimal volatile anesthetics and we will be able to prevent the use of large amounts of volatile anesthetics., It will be determined how much reduction in alveolar concentration is required in cases combined with TEA.

Nowadays, with the development of reliable anesthesia machines, "low-flow anesthesia" (LFA) is becoming more widespread, and its benefits on patient health, economy and ecology have been demonstrated. In LFA, the depth of anesthesia should not be too superficial or too deep during the time the alveolar concentration of volatile agent reaches equilibrium. Therefore, alveolar concentrations of volatile anesthetics are monitored in modern anesthesia machines. Some machines may also adjust the depth of anesthesia according to the alveolar concentration of the agent.

ELIGIBILITY:
Inclusion Criteria:

* undergoing major abdominal surgery
* Patients who will not undergoing operation for thoracic cavity
* Body Mass Index (BMI) between 20-30

Exclusion Criteria:

* denial of patients
* contraindications for thoracic epidural anesthesia
* patients who are FEV1/FVC < 60
* patients with thoracic and lomber vertebrae surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
End tidal volatile anesthetic concentration | up to 20 minutes
  End tidal volatile anesthetic concentration that keeps entropy in normal limits

SECONDARY OUTCOMES:
Total volatile anesthetic consumption | up to 2 hours
  Amount of total inhalation anesthetic consumed during surgery
Time to reach target concentration | up to 10 minutes
  Time to reach the end tidal anesthetic concentration that we set
Inhalation anesthetic amount the target concentration reached ( in the period of reaching the set alveolar concentration) | up to 5 minutes
  The amount of inhalation anesthetic consumed until reaching the target concentration
The amount of propofol | 2 minutes
  The amount of using propofol for anesthesia induction

OTHER OUTCOMES:
Total remifentanil consumption | up to end of the operation
  Total remifentanil consumption when pain index (SPI) is above normal

CONTACTS AND LOCATIONS:
Overall Officials: Nuzhet Mert Shenturk, MD, Prof, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology
Locations (1):
- İstanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD of cases included into the study will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting with the finalisation of the study ; for the next 5 years
Access Criteria: Will be determined by the institutional ethical committee

REFERENCES:
- See also: Epidural lidocaine decreases sevoflurane requirement for adequate depth of anesthesia as measured by the BIS monitor — https://www.ncbi.nlm.nih.gov/pubmed/11388531
- See also: Comparison of the effects of thoracic and lumbar epidural anesthesia on induction and maintenance doses of propofol during total i.v. anesthesia — https://www.ncbi.nlm.nih.gov/pubmed/18534970